CLINICAL TRIAL: NCT05428813
Title: The Effect of Art on Premenstrual Syndrome Symptoms: A Randomized Controlled Study
Brief Title: The Effect of Art on Premenstrual Syndrome Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Elif TUGCE CITIL, Assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-41997688-050.99-40210
Record Dates: First submitted 2022-06-09; First posted 2022-06-23 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome, Art, Women Health
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The group to which art therapy techniques will be applied.
  Interventions: Behavioral: art therapy techniques
- Control (No Intervention): The group that will continue their routine coping habits related to premenstrual syndrome.

INTERVENTIONS:
Behavioral: art therapy techniques — Art therapy is a method that allows individuals to increase their self-awareness and realize their emotions better through artistic techniques.
  Arms: Experimental

SUMMARY:
This study will be conducted to determine the effect of art therapy techniques on premenstrual syndrome symptoms.The study is a randomized controlled type study. The study will be conducted with 70 female students with premenstrual syndrome. In the study, which consists of two groups, experimental (n=35) and control (n=35), art therapy techniques will be applied to the students in the experimental group for 8 weeks. The control group will continue their routine coping habits. Both groups will be evaluated with the Premenstrual Syndrome scale at the end of the study, and the difference between the groups will be examined.

DETAILED DESCRIPTION:
First of all, ethics committee approval will be obtained by applying to the Non-Interventional Ethics Committee of the Rectorate of Kütahya Health Sciences University for the research. Then, written permission will be obtained from the Dean of the Faculty of Health Sciences of Kütahya Health Sciences University and the Department of Midwifery. In addition, written consent was obtained for the PMSS to be used in the research. At the first stage, the researcher will apply the research forms to all midwifery students willing to participate in the study without using any sampling method. The forms will be applied to volunteer and willing students after the lesson, in an appropriate classroom, by explaining the research and purpose. It is anticipated that the filling time of the forms will be 15-20 minutes on average. Then, all data will be evaluated in the SPSS program and randomization will be provided among the students who meet the inclusion criteria. Participants will be evaluated in two groups. One of the groups is the study group, where artistic techniques will be applied, and the other group is the control group, which will continue their routine coping habits for PMS. Participants will be randomly assigned to one of two groups using the www.randomizer.org program. Students in the study group (35) will do group work that will last for 30-35 minutes, one day a week, for 8 weeks, with the Artistic Techniques Education Directive prepared by the researcher holding a certificate on artistic techniques in parallel with the education they received. There is no intervention or therapy involved here. Art is used as an expressive technique, and these techniques enable students to better understand and interpret their own emotions at the end of their activity. The researcher will only apply the techniques and pose non-directive questions. At the same time, these techniques raise awareness. At the end of 8 weeks, students will be reassessed with PMSS. Students in the control group (35) will not be subjected to any application, and in parallel with the study group, they will be told to continue their routine habits regarding PMS. At the end of 8 weeks, students will be reassessed with PMSS.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Willing and volunteering to work,
* Being able to read and write and understand what one reads,
* Getting a score of 110 and above in PMSS

Exclusion Criteria:

* Engaging in any artistic activity,
* Having experienced changes in the menstrual cycle in the last 6 months

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study will be conducted with female students with premenstrual syndrome.
Enrollment: 72 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Techniques to be applied in the experimental group | It includes an 8-week process.
  At the end of 8 weeks, improvement in premenstrual syndrome symptoms is expected in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tuğçe ÇİTİL, PhD, Principal Investigator — Kütahya Health Science University
Locations (1):
- Kütahya Health Science University, Kütahya, Turkey (Türkiye)